CLINICAL TRIAL: NCT03386175
Title: Efficiency of Negative Pression Therapy With Instillation in the Debridement of Wound
Acronym: TPN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.054; 2017-A00742-51 (Other: ID RCB)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: therapy with negative pression and instillation — therapy with negative pression and instillation

SUMMARY:
the aim of the study is to evaluate the efficiency of the therapy with negative pression (TPN) and instillation in the debridement of chronic wound

DETAILED DESCRIPTION:
it is an observation study with only the aim to evaluate the percentage of fibrin before and after the specific treatment of TPN

ELIGIBILITY:
Inclusion Criteria:

* wound with debridement

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with wound and fibrin more than 70%
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-12-03 (Estimated); Study Completion 2020-12-03 (Estimated)

PRIMARY OUTCOMES:
percentage of fibrine | 1 day
  percentage of fibrine

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University hospital, Grenoble, France